CLINICAL TRIAL: NCT00895180
Title: An Open Label, Phase 2 Study Evaluating the Safety and Efficacy of IMC-3G3 or IMC-1121B in Patients With Recurrent Glioblastoma Multiforme
Brief Title: Ramucirumab or Anti-PDGFR Alpha Monoclonal Antibody IMC-3G3 in Treating Patients With Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABTC-0901 CDR0000641230; U01CA137443 (NIH); ABTC-0901; IMCL-CP-19-0801
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-11

CONDITIONS: Adult Glioblastoma Multiforme
Keywords: recurrent adult brain tumor; adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Gliosarcoma | interventions — olaratumab; Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Patients receive ramucirumab IV over 1 hour on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: ramucirumab
- Group 2 (Experimental): Patients receive olaratumab IV over 60-90 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: olaratumab

INTERVENTIONS:
Biological: olaratumab — Given IV
  Other Names: anti-PDGFR alpha monoclonal antibody; IMC-3G3
  Arms: Group 2
Biological: ramucirumab — Given IV
  Arms: Group 1

SUMMARY:
RATIONALE: Monoclonal antibodies, such as ramucirumab and anti-PDGFR alpha monoclonal antibody IMC-3G3 (Olaratumab), can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them.

PURPOSE: This phase II trial is studying how well ramucirumab or anti-PDGFR alpha monoclonal antibody IMC-3G3 works in treating patients with recurrent glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the progression-free survival rate at 6 months after treatment with ramucirumab or anti-PDGFR alpha monoclonal antibody IMC-3G3 in patients with recurrent glioblastoma multiforme.

Secondary

* To evaluate the acute and late toxicities associated with these regimens.
* To assess the objective tumor response rate.
* To estimate the overall survival of these patients.
* To describe the pharmacokinetic and pharmacodynamic profiles and immunogenicity of these regimens.

OUTLINE: This is a multicenter study. Patients are sequentially assigned to 1 of 2 treatment groups.

* Group 1: Patients receive ramucirumab IV over 1 hour on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
* Group 2: Patients receive anti-PDGFR alpha monoclonal antibody IMC-3G3 IV over 60-90 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed supratentorial glioblastoma multiforme (GBM)

  * Patients with prior low-grade glioma who progressed after radiotherapy ± chemotherapy and are biopsied and found to have GBM are eligible
* Progressive or recurrent disease after radiotherapy ± chemotherapy
* Measurable disease by contrast-enhanced MRI or CT scan

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Life expectancy ≥ 3 months
* Absolute neutrophil count ≥ 1,500/millimeter cubed (mm³)
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 gram/deciliter (g/dL)
* Creatinine ≤ 1.5 milligram/deciliter (mg/dL) OR creatinine clearance > 60 mL/min
* Total bilirubin ≤ 1.5 mg/dL
* Transaminases ≤ 3 times upper limit of normal (ULN)
* Urine protein ≤ 2+ by dipstick or urinalysis or ≤ 1,000 mg by 24-hour urine collection
* International Normalized Ratio (INR) ≤ 1.5
* Partial Thromboplastin Time (PTT) ≤ 5 seconds above ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 12 weeks after completion of study treatment
* Mini Mental State Exam score ≥ 15
* Able to undergo magnetic resonance imaging (MRI) (i.e., no pacemaker, aneurysm clip, or claustrophobia)
* No concurrent serious infection or medical illness that would jeopardize the ability of the patient to receive the treatment outlined in this study with reasonable safety including, but not limited to, any of the following:

  * Uncontrolled hypertension
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situation that would limit compliance with study requirements
* No other malignancy within the past 5 years, except curatively treated carcinoma in situ or basal cell carcinoma of the skin
* No major bleeding episode within the past 3 months
* No myocardial infarction, unstable angina pectoris, cerebrovascular accident, or transient ischemic attack within the past 6 months
* No serious or non-healing wound, ulcer, or bone fracture
* No uncontrolled or poorly controlled hypertension, despite standard medical management
* No known allergy to any of the treatment components
* No known HIV positivity or AIDS-related illness
* No uncontrolled thrombotic or hemorrhagic disorders
* No grade 3-4 gastrointestinal bleeding within the past 3 months
* No gross hemoptysis (≥ ½ teaspoon) within the past 2 months

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* At least 3 months since prior radiotherapy
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* At least 2 weeks since prior FDA-approved, non-cytotoxic agents (e.g., celecoxib, thalidomide)
* At least 3 weeks since prior investigational, non-cytotoxic agents
* More than 28 days since prior major surgery, including brain biopsy
* More than 7 days since prior subcutaneous venous access device placement
* No prior treatment with other agents that directly inhibit Platelet-Derived Growth Factor Receptor (PDGFR)α/β, Platelet-Derived Growth Factor (PDGF), Vascular Endothelial Growth Factor (VEGF), or Vascular Endothelial Growth Factor Receptor (VEGFR)s
* No concurrent therapeutic anticoagulation, chronic daily treatment with aspirin (> 325 mg/day), or other known inhibitors of platelet function
* No concurrent prophylactic hematopoietic growth factors (e.g., erythropoietin, Granulocyte Colony Stimulating Factor (G-CSF), Granulocyte-macrophage Colony Stimulating Factor (GM-CSF), or Interleukin (IL-11) during the first course of treatment
* No concurrent elective or planned surgery
* No other concurrent therapy for the tumor (e.g., chemotherapy or investigational agents)

  * Concurrent steroids allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-07; Primary Completion 2012-06-22 (Actual); Study Completion 2014-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaishri O. Blakeley, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (11):
- United States (11):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - University of California San Francisco Medical Center, San Francisco, California
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The completers include those participants with progressive disease (PD) or those who died.
Groups:
- Group 1 Ramucirumab: Participants receive ramucirumab intravenously (IV) over 1 hour on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
- Group 2 Olaratumab: Participants receive olaratumab IV over 60-90 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Group 1 Ramucirumab | Group 2 Olaratumab
Started | 40 | 40
Received at Least 1 Dose of Study Drug | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1 Ramucirumab: Participants receive ramucirumab IV over 1 hour on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Group 1 Ramucirumab | Group 2 Olaratumab | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (12.29) | 51.6 (11.81) | 51.5 (11.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 28
  Male | 28 | 24 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 39 | 38 | 77
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 38 | 37 | 75
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Progression-Free Survival Rate at 6 Months (PFS-6)
Description: PFS was defined as the start of treatment to the earliest date of tumor progression or death from any cause based on the modified Response Assessment in Neuro-Oncology Group through the American Society of Clinical Oncology (RANO) criteria. Progression is defined by any of the following: ≥ 25% increase in sum of the products of perpendicular diameters of enhancing lesions; any new lesion; or clinical deterioration. RANO is a standardized response criteria using bi-dimensional measurements of the largest contrast-enhancing area (Macdonald, 1990).
Time Frame: Start of treatment to PD or Death Up To 6 Months
Population: All enrolled participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 Ramucirumab | Group 2 Olaratumab
Number analyzed (Participants) | 40 | 40
percentage of participants | 12.5 | 7.5

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events as Assessed by NCI CTCAE v4.0 (National Cancer Institute-Common Terminology Criteria for Adverse Events)
Description: The number of participants who experienced serious adverse events (SAEs) that were considered to be related to ramucirumab or olaratumab. A summary of other non-serious adverse events and all serious adverse events, regardless of causality, is located in the Reported Adverse Events Section.
Time Frame: Start of Treatment to End of Study (Up to 13 Months)
Population: All enrolled participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Group 1 Ramucirumab | Group 2 Olaratumab
Number analyzed (Participants) | 40 | 40
participants
  SAE | 13 | 14
  Other adverse events (AEs) | 38 | 39

3. Secondary Outcome: Percentage of Participants (Pts) With Complete Response (CR), Partial Response (PR) and Minor Response (MR) (Objective Response Rate [ORR])
Description: The pts achievement of both measurement and confirmation criteria for a status of CR, PR or MR based on the modified RANO criteria.CR requires all of the following:complete disappearance of all enhancing measurable and non-measurable disease sustained for at least 4 weeks (wks);no new lesions;no corticosteroids;and stable or improved clinically.PR requires all of the following:≥ 50% decrease compared with baseline in the sum of products of perpendicular diameters of all measurable enhancing lesions sustained for at least 4 wks;no new lesions;stable or reduced corticosteroid dose;and stable or improved clinically.MR requires ≥ 25% reduction in sum of products of the perpendicular diameters of all measureable enhancing lesions sustained for at least 4 wks and no new lesions or progression of non-measurable lesions. PD is defined by any of these: ≥ 25% increase in sum of the products of perpendicular diameters of enhancing lesions;any new lesion;or clinical deterioration.
Time Frame: Start of Treatment to PD Up To 20 Months
Population: All enrolled participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 Ramucirumab | Group 2 Olaratumab
Number analyzed (Participants) | 40 | 40
percentage of participants | 0 | 2.5

4. Secondary Outcome: Median Overall Survival (OS)
Description: OS is the time from the start of treatment to the date of death. Participants who had not expired by the data analysis cutoff date were censored at their last date known to be alive.
Time Frame: Start of Treatment to Death Up To 27 Months
Population: All enrolled participants who received at least one dose of study drug. Participants censored in ramucirumab = 4 and olaratumab = 4.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Group 1 Ramucirumab | Group 2 Olaratumab
Number analyzed (Participants) | 40 | 40
Weeks | 49.5 [31.1 to 58.7] | 34.3 [24.1 to 46.9]

5. Secondary Outcome: Pharmacokinetics (PK): Concentration Maximum (Cmax) and Concentration Minimum (Cmin) of Ramucirumab
Time Frame: Cycle 7, Day 1: Prior to Infusion,1 hour (hr) Post Infusion
Population: All enrolled participants who received at least one dose of ramucirumab and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (μg/mL)
Arm/Group | Group 1 Ramucirumab
Number analyzed (Participants) | 6
microgram/milliliter (μg/mL)
  Cmin (n=5) | 85.0 (25)
  Cmax (n=6) | 396 (30)

6. Secondary Outcome: PK: Cmax and Cmin of Olaratumab
Time Frame: Cycle 3, Day 1: Prior to Infusion, 1 hr Post Infusion
Population: All enrolled participants who received at least one dose of Olaratumab and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Group 2 Olaratumab
Number analyzed (Participants) | 5
μg/mL
  Cmin (n=5) | 145 (22)
  Cmax (n=5) | 515 (23)

7. Secondary Outcome: Pharmacodynamics (PD) Profiles
Time Frame: Cycle 7, Day 1: Prior to Infusion, 1 hr Post Infusion
Population: Zero participants were analyzed for pharmacodynamic profile as the plasma collection procedure in this study was not fit for this purpose.
Arm/Group | Group 1 Ramucirumab | Group 2 Olaratumab
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Percentage of Participants With Anti-Olaratumab Antibodies (ADA)
Description: Percentage of Participants with Treatment Emergent (TE) anti-olaratumab antibodies were participants with a 4-fold increase (2 dilutions) increase over a positive baseline antibody titer or for a negative baseline titer, a participant with an increase from the baseline to a level of 1:20.
Time Frame: Start of Treatment to 30-day Post Infusion Follow Up (Up to 6 Months)
Population: All enrolled participant who had any amount of olaratumab and evaluable anti-olaratumab antibody data.
Measure: Number; unit: percentage of participants
Arm/Group | Group 2 Olaratumab
Number analyzed (Participants) | 26
percentage of participants | 0

9. Secondary Outcome: Percentage of Participants With Anti-Ramucirumab Antibodies (ADA)
Description: Percentage of Participants with Treatment Emergent (TE) anti-ramucirumab antibodies were participants with a 4-fold increase (2 dilutions) increase over a positive baseline antibody titer or for a negative baseline titer, a participant with an increase from the baseline to a level of 1:20.
Time Frame: Start of Treatment to 30-day Post Infusion Follow Up (Up to 6 Months)
Population: All enrolled participants who had any amount of ramucirumab and evaluable anti-ramucirumab antibodies.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 Ramucirumab
Number analyzed (Participants) | 32
percentage of participants | 3.1

ADVERSE EVENTS:
Arm/Group | Group 1 Ramucirumab | Group 2 Olaratumab
Serious Adverse Events (participants affected / at risk) | 13/40 | 14/40
Other Adverse Events (participants affected / at risk) | 38/40 | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Ramucirumab (N=40) | Group 2 Olaratumab (N=40)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Shunt infection (Infections and infestations) | 0 (0) | 1 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incorrect storage of drug (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Brain edema (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral hematoma (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 3 (3) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hemorrhage intracranial (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Vasogenic cerebral edema (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Group 1 Ramucirumab (N=40) | Group 2 Olaratumab (N=40)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
Cushingoid (Endocrine disorders) | 4 (4) | 2 (2)
Vision blurred (Eye disorders) | 3 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 5 (7) | 10 (17)
Faecal incontinence (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (9) | 12 (20)
Vomiting (Gastrointestinal disorders) | 5 (5) | 7 (9)
Asthenia (General disorders) | 3 (3) | 1 (1)
Chills (General disorders) | 2 (2) | 3 (3)
Fatigue (General disorders) | 19 (25) | 18 (24)
Gait disturbance (General disorders) | 6 (10) | 6 (7)
Non-cardiac chest pain (General disorders) | 2 (2) | 3 (3)
Edema peripheral (General disorders) | 6 (8) | 5 (6)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (5) | 2 (2)
Vaginal infection (Infections and infestations) | 1/12 (2) | 0/16 (0)
Contusion (Injury, poisoning and procedural complications) | 6 (7) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 6 (9) | 4 (4)
Weight increased (Investigations) | 2 (2) | 4 (5)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 3 (7) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 3 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Aphasia (Nervous system disorders) | 6 (9) | 5 (6)
Balance disorder (Nervous system disorders) | 3 (3) | 2 (2)
Cognitive disorder (Nervous system disorders) | 5 (7) | 1 (1)
Convulsion (Nervous system disorders) | 5 (6) | 4 (9)
Disturbance in attention (Nervous system disorders) | 3 (4) | 0 (0)
Dizziness (Nervous system disorders) | 5 (5) | 8 (9)
Dysarthria (Nervous system disorders) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 16 (21) | 12 (20)
Hemiparesis (Nervous system disorders) | 1 (1) | 4 (7)
Hypoesthesia (Nervous system disorders) | 3 (4) | 1 (1)
Memory impairment (Nervous system disorders) | 3 (3) | 4 (4)
Tremor (Nervous system disorders) | 4 (5) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (2)
Confusional state (Psychiatric disorders) | 6 (7) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (2) | 8 (8)
Proteinuria (Renal and urinary disorders) | 0 (0) | 5 (10)
Urinary incontinence (Renal and urinary disorders) | 1 (2) | 3 (3)
Amenorrhea (Reproductive system and breast disorders) | 0/12 (0) | 1/16 (1)
Dysmenorrhea (Reproductive system and breast disorders) | 1/12 (1) | 0/16 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (8)
Hypertension (Vascular disorders) | 2 (3) | 10 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the ABTC publication, JHU will submit the draft of any proposed publication to ImClone at least thirty (30) days prior to submission for publication and agrees to withhold any such submission for an additional period, not to exceed ninety (90) days to allow ImClone to file patent applications. If Confidential Information is in the publication, it will notify JHU, which will insure such Confidential Information is redacted.